CLINICAL TRIAL: NCT04389138
Title: Is Physiotherapy Effective for People With Early Parkinson's (PEEP) a Feasibility Study
Brief Title: Is Remote Physiotherapy Effective for People With Early Parkinson's (PEEP)
Acronym: PEEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DHRD/2018/104
Record Dates: First submitted 2020-04-28; First posted 2020-05-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparison (No Intervention): In this arm participants will attend 3 study visits to complete study questionnaire and assessments. In between these visits, participants will be asked to wear an activity monitor and record an activity diary for one week. Other than this, participants will continue to receive only standard of care treatment.
- Intervention arm (Experimental): In this arm participants will attend the same 3 study visits to complete study questionnaires and assessments. Participants will be asked to wear an acitvity monitor and record an activity diary for one week after the study visits. In between baseline and 6 month follow up, intervention arm participants will receive study physiotherapy. This will consist of an individual assessment and 4 additional sessions of physiotherapy.
  Interventions: Other: Physiotherapy Intervention

INTERVENTIONS:
Other: Physiotherapy Intervention — Physiotherapy intervention will include an assessment to identify individual areas that physiotherapy should target. Intervention will be based on the core areas recommended by the European Physiotherapy Guideline for Parkinson's Disease: physical capacity (muscle power, tone, joint range of movement, exercise tolerance and pain), transfers, manual dexterity, balance and gait. Posture is incorporated as part of these 5 core areas. The intervention will be delivered over 4 visits.
  Arms: Intervention arm

SUMMARY:
Parkinson's disease is a progressive neurodegenerative condition affecting 145,500 people in the UK. The condition impairs movement leading to gait and dexterity problems. Various types of exercise are beneficial for both motor and non-motor symptoms such as depression.

The World Health Organisation's (WHO) recommendations on exercise include at least 150 minutes of moderate-intensity aerobic physical activity per week . People with Parkinson's may struggle to achieve this because of movement problems and fatigue. Physiotherapists may have a role in persuading people to exercise and supporting them in their activity goals. While studies show that Parkinson's patients with falls or gait freezing clearly benefit form physiotherapy, there is at present no robust evidence to demonstrate the impact of physiotherapy early in the course of the illness.

PEEP seeks to explore the effectiveness of physiotherapy for early Parkinson's (ie within 4 years of diagnosis and before onset of falls).

It comprises three distinct parts:

1. A survey of people with Parkinson's exploring their experience and opinions with respect to physiotherapy for early Parkinson's
2. A feasibility randomised controlled trial (fRCT)
3. A qualitative process evaluation. The fRCT will aim to recruit and randomise 40 people withParkinson's who have been diagnosed in the last 4 years and have had no physiotherapy. These participants will undergo several assessments at baseline, 3 months and 6 months, and will also have 7 days' worth of activity monitoring done via physical diary and a commercially available activity tracker to determine levels of activity. Participants randomised to the intervention arm will also receive 5 physiotherapy sessions (1 for assessment and 4 for treatment) additional to standard NHS care.

Staff and some participants involved in the fRCT will be included in a qualitative process evaluation to assess the acceptability and feasibility of the intervention and the research assessments.

DETAILED DESCRIPTION:
The Principle research question is:

* To explore the experience and opinions of people with Parkinson's in relation to physiotherapy and exercise in early disease.
* To develop a physiotherapy exercise intervention for people with early Parkinson's disease using insights from patients and professionals.
* To explore the feasibility of a future definitive randomised controlled trial, which would investigate the clinical and cost effectiveness of the physiotherapy intervention

The project has 3 elements:

1. A survey of people with Parkinson's exploring their views about physiotherapy and exercise.
2. A feasibility randomised trial of Parkinson's versus usual care for people with Parkinson's.
3. A qualitative process evaluation exploring view of participants, research nurses and treating physiotherapists on the acceptability and of the intervention and the research assessments.

Survey of people with Parkinson's:

Online and paper survey will be available for people with Parkinson's to complete. The survey will be posted on the Parkinson's UK website. The survey will be open to UK residents with Parkinson's who have been diagnosed within the last 4 years.

Feasibility Randomised Controlled Trial The project will also consist of a Feasibility trial of physiotherapy for early Parkinson's versus usual care. Randomised controlled trial. Blinded assessment of outcomes. Parallel group design. Patient will be followed up at 3 and 6 months after the baseline visit. The RCT will be set in two NHS tertiary care centres.

At baseline, the following study procedures will be completed. Eligibity assessment by the PI or delegated research team member. 1. Demographics, medical history, medication history, physical examination (DOB, Height, Weight, Sex) The following Standard Questionnaires will be completed at the baseline visit.

* Montreal cognitive assessment (MoCA). This is a measure of cognition widely used in Parkinson's clinics (38).
* PDQ-39.
* UPDRS. This is a Parkinson's assessment tool that includes subsections looking at motor symptoms and signs, non-motor symptoms, activities of daily living and mood.
* SF-12. This is a measure of health related quality of life. Where the participant with Parkinson's has a carer who has agreed to take part in the study the investigator will ask the carer to complete this assessment.
* LPAS
* Mini-BEST
* Tragus to wall distance. Activity diaries: Participants will be given an activity diary and asked to record their activity over the next 7 days (starting the day after the initial visit). The activity diary will be returned to the research team in a pre-paid addressed envelope that will be provided to the participant.

Activity monitors: The research nurse will provide each participant with a activity monitor and provide instruction on how to use and charge at home. The monitor will be provided fully charged. The device will be worn on the wrist. Participants will be asked to wear the device for the next 7 days. The device can be worn while showering or swimming. The device should then be returned to the research team in a stamped addressed envelope provided, along with the completed activity diary. The main outcomes of interest from the activity monitors will be average daily step count and active minutes/day.

For Participants randomised to the intervention arm, they will attend an initial assessment visit followed by 4 physiotherapy intervention visits. At each of these 5 visits, a checklist will be completed by the physiotherapist to document what has been delivered as part of the intervention.

The following assessments will take place at 3 months and 6 months after baseline visit.

* Medication history.
* PDQ-39
* SF-12
* Number of falls
* 7 day activity diary
* Activity monitor (7days)
* LPAS
* Tragus to wall
* Record of outside of study therapy interventions.
* Adverse event register
* The outcome assessor will be asked if they have been unblinded.
* The mini-BEST will be measured at 3 months.

Qualitative Process evaluation.

Both staff and participants will be interviewed to explore views on care and the intervention. Interviews will last roughly 1 hour. Interviews will include:

* 6-10 physiotherapists
* 6-8 Participants from the Randomised controlled trial
* 2-4 Research Nurses from the Randomised controlled trial.

ELIGIBILITY:
INCLUSION CRITERIA Survey of people with Parkinson's

* People with Parkinson's aged >18, diagnosed within the last 4 years.
* Able to read and write English.
* Willing to take part in survey.

Feasibility RCT

* Parkinson's disease diagnosed <4 years before study entry
* Parkinson's diagnoses fits UK Brain Bank criteria
* Age ≥18 years at study entry
* Willingness to attend for physiotherapy interventions
* Ability to transfer and walk independently
* Stable Parkinson's medication:
* Parkinson's medication not commenced or altered in last 2 months.
* Changes to Parkinson's medication are not planned/scheduled in next 6 months
* Participants not on PD medication can be recruited. (Treating clinicians can change Parkinson's medication during study according to clinical need and changes will be recorded on case report form.)

Qualitative process evaluation

* Participants of the feasibility RCT
* Physiotherapists within the trial conducting assessments and treatments.
* Research Nurses who delivered the RCT

EXCLUSION CRITERIA

* Hoehn-Yahr stage 4-5 (Hoehn -Yahr staging included as Appendix 2)
* Lacks capacity to consent
* Meets the criteria for commencement of the Gold Standards Framework (see Appendix 3)
* Falls [more than 1 fall in the 3 months prior to enrolment]
* Freezing of gait
* Already had outpatient (OP) or community physiotherapy for Parkinson's:

OP physiotherapy for trauma or arthritis will not be exclusion A single one -off assessment of Parkinson's by a physiotherapist will not be an exclusion Attendance at exercise classes which are not supervised by a physiotherapist will not count as an exclusion.

IP physiotherapy will not count as an exclusion Unable to communicate in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Number of Eligible Patients | Collected up to 104 weeks.
  Screening data will be collected to understand how many participants are eligible for the study. This data is a feasibility outcome which will be used to determine if a larger scale definitive study is possible. The data collected surrounding number of eligible patients can help to power in any future study.
Length of waiting time from enrolment to delivery of intervention. | Collected up to 130 weeks.
  Measurement of time between consent and the completion of the physiotherapy intervention. This will be considered a feasibility outcome to determine whether the intervention is feasible for a larger definitive study.
Change from baseline to follow up time points for all clinical outcomes | Collected up to 130 weeks.
  The change in all clinical outcomes from baseline to 6 months, the standard deviation, and the effect size of clinical outcomes to define the primary outcome for a future definitive trial.
Completeness of data collection for clinical outcomes. | Collected up to 130 weeks.
  Percentage of data completeness will be collected as a feasibility outcome to determine if clinical outcomes can be used in a definitive study
Adherence of clinical staff to intervention protocol. | Collected up to 130 weeks
  This outcome will assess whether the planned number of physiotherapy treatment sessions (4) and follow up telephone consultations (2) are undertaken. A bespoke checklist will be used to document each phone call and physiotherapy visit to outline that the intervention has been delivered.
Whether the person assessing the clinical outcomes at baseline, 3 month and 6 month outcomes is blinded | Collected up to 130 weeks.
  This will be self reported by the clinician to indicate if the blind was broken. This will be used as a feasibility outcome to determine if any future definitive study can be blinded
Feasibility of Using Activity Monitor | Collected up to 130 weeks.
  • Practicalities (including time taken to retrieve and record data) of using commercially available activity monitors as an outcome measure.
Feasibility and Acceptability of Study Intervention through Qualitative interviews with staff and Clinicians working on study. | Collect
  Interviews will cover the following topics to assist in determining if a definitive future trial is feasible.
  * The different elements of usual care in two centres, including use of physiotherapy.
  * Time needed for research nurse to complete and record all study assessments and outcomes as assessed by qualitative interview.
  * Recruitment rate. Describe reasons patients chose not take part.
  * Feedback from the clinicians delivering the intervention about which elements of the intervention could be delivered in a large RCT, the optimal number of patient-therapist interactions and appropriateness of outcomes.
  * Delivery of the proposed intervention by the physiotherapy services at baseline assessment, follow up visits, telephone reviews.
Feasibility and Acceptability of Study Intervention through Qualitative interviews with participants who participated in the study. | Collected up to 130 weeks
  Purpose of the interviews is to determine if a future definitive trial is feasible and acceptable for participants. Interviews will cover the following topics.
  * Patient adherence to visit and treatment schedule. Facilitators and barriers for attending the visits and undertaking the required treatment.
  * Feedback from the patients about the acceptability of the treatment programme and the study assessments.

SECONDARY OUTCOMES:
Parkinson's Disease Questionnaire 39 (PDQ-39) | Collected at Baseline, 3 and 6 month follow up
  Clinical Outcome collected by Questionnaire. Scored 0-100, 100 is considered the worst outcome.
Unified Parkinson's Disease Rating Scale (UPDRS) | Collected at Baseline, 3 and 6 month follow up
  a global measure of Parkinson's severity that includes subsections looking at motor symptoms and signs, non-motor symptoms, activities of daily living and mood. Lower scores better. 4 subscales: non-motor 0-52, motor experience0-52, motor examination 0-132, motor complication 0-24.
Activity | Collected up to 6 months.
  Activity as captured using Activity diaries: types of activity; total number of minutes per day and per week at different levels of perceived exertion based on Borg scale 620.
Activity Monitor Data | Collected up to 6 months.
  Step count, minutes of sleep (Rem, light, deep) and very & moderately active minutes using Fitbit Inspire HR activity monitors
Short Form 12 (SF12) | Collected at baseline, 3 and 6 month follow up visit
  measuring carer well-being, where a carer is available. Higher scores are better (Better health status). 50 is average score. 40-60 is range within 1 standard deviation of mean score. Scores 30-70 represent scores within 2 standard deviations of mean. There are subscales for Physical health and mental health.
Lindop Parkinson's Assessment Scale [LPAS] | Collected at baseline, 3 and 6 month follow up visit
  Assessment of Gait (LPAS includes Timed up and Go) and transfers (timed bed transfers - included in LPAS)
Mini Balance Evaluation Systems Test (mini-BEST) | Collected at baseline, 3 and 6 month follow up visits
  Questionnaire assessment
Tragus to Wall distance (posture assessment) | Collected at baseline, 3 and 6 month follow up visits
  posture assessment. 10 cm - 12cm range is considered the better range. Higher scores up to 30cm in rare cases suggest worse health outcomes.
Number of Falls | Collected at baseline , 3 month and 6 month follow up visits.
  Self reported outcome

CONTACTS AND LOCATIONS:
Overall Officials: Robert Skelly, Principal Investigator — University Hospitals of Derby and Burton NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No